CLINICAL TRIAL: NCT01908946
Title: Automated SMS Reminders to Parents on Their Cell Phones Can Significantly Improve the on Time Vaccination Rates Among Children in Pakistan
Brief Title: Automated SMS Reminders to Parents on Their Cell Phones Can Significantly Improve the on Time Vaccination Rates Children in Pakistan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aga Khan University (Other)
Collaborators: World Health Organization (Other)
Responsible Party: Principal Investigator, Dr Abdul Momin Kazi, Senior Instructor, Aga Khan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: EM-2013-IER-RPC-TSA-008
Record Dates: First submitted 2013-07-15; First posted 2013-07-26 (Estimated); Last update posted 2013-07-26 (Estimated); Status verified 2013-07

CONDITIONS: Vaccination Failure
Keywords: Polio
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SMS Reminders (Experimental): SMS reminders
  Interventions: Behavioral: SMS reminders
- Standard verbal counseling (No Intervention): One time standard verbal counseling at the time of initial visit and timing for EPI vaccines at 6, 10 and 14 weeks

INTERVENTIONS:
Behavioral: SMS reminders — SMS reminders for vaccination visit at 6, 10 and 14 weeks of life.
  Arms: SMS Reminders

SUMMARY:
The investigators plan to test the effectiveness of reminders to parents/guardians on cell phones through short messaging system (SMS) in improving the on-time routine immunization for children in Pakistan. SMS message as a reminder tool can be very effective in health care settings at public health scale. This study will be conducted in an urban- squatter settlement area, Ibrahim Haidry union council in Karachi. Parents/guardians of children randomized in intervention arm will be sent SMS reminders vaccination visit reminders at 6, 10 and 14 weeks of life.

DETAILED DESCRIPTION:
The immunization coverage in Pakistan is still well below the desired level, leading to continued polio transmission, large measles outbreaks and thousands of deaths from vaccine-preventable illnesses. A major reason for poor childhood vaccine coverage is the lack of awareness among parents regarding the need for immunization in children, and the importance of completing the entire series of vaccines. This result in significant drop-out between vaccines delivered at birth and later in the infancy period. Customized short messaging system (SMS) text can be designed as personally tailored messages to remind and inquire parents regarding vaccination for their children according to the EPI schedule. We plan to test the effectiveness of reminders to parents/guardians on cell phones through short messaging system (SMS) in improving the on-time routine immunization for children in Pakistan. This study will be conducted in an urban- squatter settlement area, Ibrahim Haidry union council in Karachi, Pakistan. Our experimental plan has three components: First, we will conduct baseline survey of parents at our study site to explore their preferences for text for immunization reminders. Simultaneously, we will develop a computerized application for reminders scheduling. This application will contain the phone number, message information, language preferences and date on which the message will be sent. It will be interfaced with the gateway to send the message. Lastly, we will conduct a randomized controlled trial to determine the effectiveness of automated SMS reminders to parents in improving the on-time vaccination rates in children. If the result shows that the vaccines compliance can be increased through the SMS reminders, this program can be incorporated with the existing systems to collect the cell phone numbers of parents at the time of child's first contact with the health system and sending auto generated reminders for vaccine compliance at national level.

ELIGIBILITY:
Inclusion Criteria:

* Child should be less than 14 days of age
* Parent/guardian or at least one person in the household having a valid cell phone connection
* Parent/guardian provides consent

Exclusion Criteria:

* Child more than 14 days of age
* Not a valid cell phone connection in the household
* Parent/guardian not providing consent

Max Age: 14 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2013-05; Primary Completion 2013-10 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Improvement in the vaccination coverage due to SMS reminders | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ibrahim M Abdel Rahim, MBBS, Study Director — Ibrahim Mohamed ABDEL RAHIM
Locations (1):
- Aga Khan University, Karachi, Sindh, Pakistan